CLINICAL TRIAL: NCT02968446
Title: The Effect of Oral Vitamin D (Cholecalciferol) Supplementation After Topical Application With Valchlor
Brief Title: Effect of Vitamin D After Application With Valchlor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kurt Lu, Assistant Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09-16-36C; U01AR064144-01 (NIH); CASE3416 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Skin Irritation
Keywords: Valchlor; Vitamin D; Healthy Volunteer
MeSH Terms: interventions — Cholecalciferol; Amines; Mechlorethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: 4 placebo - 0 Vitamin D with Valchlor (Placebo Comparator): Participants will be given 4 placebo capsules and 0 cholecalciferol (Vitamin D) capsules after being treated with Valchlor.
  Interventions: Dietary Supplement: 4 placebo; Drug: Valchlor
- Group 2: 0 placebo - 4 Vitamin D with mechloroethamine (Experimental): Participants will be given 0 placebo capsules and 4 cholecalciferol capsules to total 200,000 IU of cholecalciferol (Vitamin D) after being treated with Valchlor.
  Interventions: Dietary Supplement: 4 Vitamin D; Drug: Valchlor

INTERVENTIONS:
Dietary Supplement: 4 placebo — subjects will take orally 4 pills without any active ingredients which are of the same size, shape and color as the study pills
  Other Names: placebo
  Arms: Group 1: 4 placebo - 0 Vitamin D with Valchlor
Dietary Supplement: 4 Vitamin D — subjects will take orally four pills for a single dose of 200,000 IU of Vitamin D (cholecalciferol)
  Other Names: cholecalciferol
  Arms: Group 2: 0 placebo - 4 Vitamin D with mechloroethamine
Drug: Valchlor — Twice during the study, subjects will be given 0.016% Valchlor at 3 locations (for a total of 6 locations) in the inner arm using Finn ChambersTM
  Other Names: Mechlorethamine

SUMMARY:
The purpose of this research study is to evaluate the effects of an oral Vitamin D on the body's immune system.

An interest has been growing because studies have shown that Vitamin D may reduce inflammation and harmful effects in the body, however, the best dose for Vitamin D is still unknown.

Inflammation is the body's physical response to infection, injury, or long term disease. Pain, redness, heat, and sometimes loss of function are all signs of inflammation in the body. This study will look at product use, testing skin irritation in healthy volunteers and seeing how Vitamin D may help stop or reduce inflammation and skin irritation, which could one day help doctors prescribe Vitamin D to patients with long term disease to relieve their symptoms.

DETAILED DESCRIPTION:
Primary Endpoint To determine the effect of a topical application of Valchlor on human subjects at the clinically approved dose.

Secondary Endpoint To establish the efficacy of cholecalciferol (vitamin D3) in reducing skin irritation 48 hours after topical application of Valchlor.

ELIGIBILITY:
Inclusion Criteria:

* Must be in general good health
* Fitzpatrick Skin Type I-VI
* Able to list all current medications and medical conditions
* Capable of giving informed consent

Exclusion Criteria:

* Women who are pregnant, nursing, or who may become pregnant in the next 3 months
* Participants taking illegal drugs
* Currently taking ketoconazole, colestipol, cholestyramine, phenobarbitol, phenytoin, or mineral oil
* Currently consuming 800IU or more of vitamin D a day
* Subjects whose BMI are > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in skin erythema | Up to 1 week after mechloroethamine exposure
  Skin erythema (redness) will be quantified using a CR300 chromameter. The difference in erythema between exposed and non-exposed skin will be calculated after valchlor exposure

SECONDARY OUTCOMES:
Change in skin thickness | Up to 1 week after mechloroethamine exposure
  Skin thickness, an acute measure of edema, was quantified using a Mitutoyo 9mm dial caliper. Thickness measurements will be repeated in triplicate and the mean was used for all calculations. The difference in thickness between exposed and non-exposed skin will be calculated after valchlor exposure.
Change in TNF-alpha expression | Up to 120 hours after mechloroethamine exposure
  A 6 mm punch biopsy specimen will be obtained from the valchlor exposure site 48hr after exposure. RNA will be extracted from fresh frozen punch biopsies using the RNeasy Lipid Mini Kit, and tissue mRNA expression of TNF-α will be quantified
Change in iNOS expression | Up to 120 hours after mechloroethamine exposure
  A 6 mm punch biopsy specimen will be obtained from the valchlor exposure site 48hr after exposure. RNA will be extracted from fresh frozen punch biopsies using the RNeasy Lipid Mini Kit, and tissue mRNA expression of iNOS will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Lu, MD, Principal Investigator — Northwestern University
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ernst MK, Evans ST, Techner JM, Rothbaum RM, Christensen LF, Onay UV, Biyashev D, Demczuk MM, Nguyen CV, Honda KS, McCormick TS, Tsoi LC, Gudjonsson JE, Cooper KD, Lu KQ. Vitamin D3 and deconvoluting a rash. JCI Insight. 2023 Jan 24;8(2):e163789. doi: 10.1172/jci.insight.163789. PMID 36692020